CLINICAL TRIAL: NCT03112317
Title: Does Mild Hypothermia Increase Intra-Operative Blood Loss and Surgical Site Infections in Major Abdominal Surgery?
Brief Title: Mild Hypothermia Influence on Patient Outcome in Major Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: University College of Southeast Norway (Other)
Responsible Party: Sponsor
Other Study IDs: REK Vest (2016/2193)
Record Dates: First submitted 2017-03-26; First posted 2017-04-13 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-02

CONDITIONS: Surgical Site Infection; Bleeding
Keywords: Surgery; Hypothermia; Prevention; Surgical Site Infection; Bleeding; Surgical instruments
MeSH Terms: conditions — Surgical Wound Infection; Hemorrhage; Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypothermia: Patients with mild hypothermia at start of the surgery
  Interventions: Other: Prevention of hypothermia
- Normothermia: Patients with normal core temperature at start of surgery.
  Interventions: Other: Prevention of hypothermia

INTERVENTIONS:
Other: Prevention of hypothermia — Patients are routinely warmed with forced air warming blankets, regular blankets, pre warmed intravenous fluid. Routines are ensured with use of the WHO Surgical Safety Checklist. The intervention is the use of operating theatre care measures to prevent mild hypothermia in surgical patients.
  Other Names: Forced air warming blankets

SUMMARY:
This study investigate associations between mild hypothermia (patients' core temperature ≤ 36.0 degrees Celsius) and intra-operative blood loss and surgical site infections (SSI) in patients undergoing major abdominal surgery.

DETAILED DESCRIPTION:
This study evaluates associations between patients' core temperature during surgery and intra-operative blood loss, and to SSI. Additionally, the investigators observe the use of hypothermia prevention measures in operating theaters, use of surgical safety checklists. SSI is registered at discharge from hospital and up to 30 days post-discharge.

The goal of the study is to contribute to focus on prevention of even mild hypothermia in surgery.

This study is of interest for healthcare personnel as operating room nurses, surgeons, nurse anaesthetists, anaesthesiologists, ward nurses, post anaesthetic care unit nurses, and other healthcare staff involved in the in-hospital surgical pathway.

ELIGIBILITY:
Inclusion Criteria:

* Patients (men or women) above 18 years, undergoing abdominal or gynecological surgery with laparotomy or laparoscopy.

Exclusion Criteria:

* Surgical procedures with intentional reduction of core temperature. Patients under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consist of patients undergoing abdominal or gynecologic laparatomy or laparoscopy in a tertiary teaching hospital in Norway.
Sampling Method: Probability Sample
Enrollment: 3059 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Intra-operative blood loss (mL) in surgical patients | Within the surgical procedure
  Bleeding that occur during the surgical procedure

SECONDARY OUTCOMES:
Peri-operative blood loss (registered by ICD-10 codes) | Within the duration of the surgical procedures, an average of 2.5 hours
  Bleeding requiring blood transfusion peri-operatively
Number of patients with Surgical Site Infections after surgery | Up to 30 days after discharge from hospital
  Post-operative surgical site infections present before discharge from hospital
Number of patients with Surgical Site Infection | Up to 30 days after discharge from hospital
  Post-operative surgical site infection present after discharge from hospital
Days admitted in hospital | Hospital stay up to 13 days on average
  Length of stay in hospital
Hours admitted in post operative care unit (PACU) | On average up to 14 hours
  Length of stay in PACU

CONTACTS AND LOCATIONS:
Overall Officials: Arvid S Haugen, PhD, MSc, Principal Investigator — Haukeland University Hospital
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen, Hordaland
  - Haukeland University Hospital, Bergen

IPD SHARING:
Plan to Share IPD: Yes
Anonymous individual data is allowed to share, thought such request must be approved by the REK West. Data will be available from the primary investigator.

REFERENCES:
- Available data/document: Study Protocol: REC West (2016-2193) — https://helseforskning.etikkom.no/komiteerogmoter/vest/sekretariat?region=10796&p_dim=34985&_ikbLanguageCode=us — Study protocol is available on request to Regional Committees for Medical and Health Research Ethics.